CLINICAL TRIAL: NCT00005827
Title: Phase I Single and Multiple-Dose Safety and Pharmacokinetic Clinical Study of Genistein in Normal Volunteers and in Prostate Neoplasia (Multiple Dose Safety and Pharmacokinetic Clinical Study of Genistein in Prostate Neoplasia)
Brief Title: Genistein in Treating Patients With Stage II, Stage III, or Stage IV Prostate Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 9711; UNC-GCRC-1203; NCI-G00-1788; CDR0000067840 (Other: PDQ number)
Record Dates: First submitted 2000-06-02; First posted 2004-04-20 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: genistein

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase I trial to determine the effectiveness of genistein in treating patients who have stage II, stage III, or stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and pharmacokinetics of genistein in patients with stage II, III, or IV prostate cancer.

OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are randomized to one of two treatment arms. Arm I: Patients receive oral genistein twice daily. Arm II: Patients receive oral placebo twice daily. Treatment continues for 3 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage B, C, or D adenocarcinoma of the prostate not amenable to surgery

PATIENT CHARACTERISTICS: Age: 40 and over Performance status: ECOG 0-2 Life expectancy: At least 6 months Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Transaminases less than 4 times upper limit of normal Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease Other: No significant abnormalities of internal organs, neurologic status, or biochemical levels No history of seizures No concurrent serious illness No acute infection requiring antibiotic therapy except chronic urinary tract infection No other prior or concurrent malignancy within the past 2 years except nonmelanoma carcinoma of the skin No history of substance abuse or addiction No alcohol intake greater than 2 drinks/day or 14 drinks/week No diet containing more than 20 mg of genistein/day No known soy intolerance No prior breast cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: At least 3 months since prior hormonal therapy OR No concurrent estrogen Other concurrent hormonal therapy allowed if stable regimen for more than 3 months Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics At least 3 weeks since prior surgery and recovered Other: At least 6 weeks since prior antibiotics No concurrent genotoxicity therapy

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-12; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Fischer, PhD, MPH, RD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina, United States